CLINICAL TRIAL: NCT00798759
Title: Examination of Ocular Surface Effects With Administration of TRAVATAN Z® and XALATAN®
Brief Title: Examination of Ocular Surface Effects With Administration of Travatan Z and XALATAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-050
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost (Experimental): One drop self-administered in the study eye(s) once daily at night for 12 weeks
  Interventions: Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®)
- Latanoprost (Active Comparator): One drop self-administered in the study eye(s) once daily at night for 12 weeks
  Interventions: Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®)

INTERVENTIONS:
Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 12 weeks (84 days). Referred to as travoprost.
  Other Names: TRAVATAN Z®
  Arms: Travoprost
Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 12 weeks (84 days). Referred to as latanoprost.
  Other Names: XALATAN®
  Arms: Latanoprost

SUMMARY:
The purpose of this study is to compare two ophthalmic solutions in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Diagnosis of open-angle glaucoma or ocular hypertension in at least one eye.
* Intraocular pressure (IOP) controlled with BAK (benzalkonium chloride) preserved IOP-lowering medication for 1 year, with last 6 months on XALATAN® monotherapy.
* Best corrected visual acuity of -0.6 logMAR or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Treatment with BAK preserved artificial tears within 30 days of Visit 1.
* Known or suspected Sjogren's disease.
* Uncontrolled IOP.
* History or evidence of infectious or inflammatory ocular conditions.
* Progressive retinal or optic nerve disease.
* Ocular laser surgery within 3 months of Visit 1.
* Keratorefractive ocular laser procedures, corneal surgery or surgery to the corneal surface within 1 year of Visit 1.
* Current use of punctal plugs or punctal cautery.
* Use of systemic medications that has not been stable for 30 days prior to Visit 1.
* Use of contact lens within 30 days of Visit 1.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 22 US study centers. Eligible patients having a diagnosis of open-angle glaucoma or ocular hypertension and on XALATAN® monotherapy for six months prior to Visit 1 were enrolled.
Pre-assignment Details: 236 patients were enrolled in the study and evaluated for safety. Baseline characteristics are presented for all patients who received test article and completed the study (intent-to-treat): 215.
Period: Overall Study
Arm/Group | Travoprost | Latanoprost
Started | 117 | 119
Completed | 109 | 106
Not Completed | 8 | 13
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 4 | 8
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost | Latanoprost | Total
Number analyzed (Participants) | 109 | 106 | 215
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (12.1) | 69.0 (10.4) | 67.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 71 | 137
  Male | 43 | 35 | 78

OUTCOME MEASURES:

1. Primary Outcome: Mean Change at 12 Weeks (Day 84) From Baseline (Day 0) in Tear Film Break-Up Time (TFBUT)
Description: Tear film break-up time was assessed by the same examiner both visits using the same slitlamp/settings. Examiner instilled fluorescein onto the patient's eye, after which the patient blinked several times, then kept the eye open. Immediately thereafter, the examiner used a stopwatch to time the occurrence of the first break in the fluorescein film. Three consecutive measurements were taken and averaged for actual TBUT. TBUT at Baseline (Day 0) was subtracted from TBUT at 12 weeks (Day 84) and reported as change. A higher number represents a lengthening in the tear film break up time.
Time Frame: Day 0, Day 84
Population: Intent-to-Treat: All patients who received test article and completed the trial.
Measure: Mean (Standard Error); unit: Seconds
Groups:
- Travoprost; Latanoprost: One drop self administered in the study eye(s) once daily at night for 12 weeks
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 109 | 105
Seconds | 0.7 (0.1) | 0.6 (0.2)

2. Secondary Outcome: Mean Change at 12 Weeks (Day 84) From Baseline (Day 0) in Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a 12-question validated questionnaire (resultant overall 0-100 score) used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision, where 0 = normal and 100 = severe. The OSDI questionnaire was administered at both visits and completed by the patient with no assistance from the office staff, physician, or anyone else. The baseline OSDI score was subtracted from the 12-week OSDI score and reported as change. A negative number represents a perceived improvement in ocular health.
Time Frame: Day 0, Day 84
Population: Intent-to-Treat: All patients who received test article and completed the trial.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 108 | 106
Units on a scale | -1.9 (1.2) | 0.6 (1.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 22 December 2008 to 20 May 2009.
Description: This reporting group includes all patients who received test article.
Arm/Group | Travoprost | Latanoprost
Serious Adverse Events (participants affected / at risk) | 1/117 | 2/119
Other Adverse Events (participants affected / at risk) | 7/117 | 3/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost (N=117) | Latanoprost (N=119)
Blood urine present (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost (N=117) | Latanoprost (N=119)
Dry Eye (Eye disorders) | 7 | 3

LIMITATIONS AND CAVEATS:
The subjective nature of the OSDI may not be sensitive enough to detect the effects of preservatives on the corneal surface. The measurement and quantification of OSD remains a considerable clinical challenge. (Pflugfelder and Baudoin, 2011)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.